CLINICAL TRIAL: NCT02596620
Title: The Efficacy of 10-day Metronidazole and Levofloxacin Containing Sequential Therapy and 10-day Levofloxacin-containing Triple Therapy In Second Line Helicobacter Pylori Eradication Therapies
Brief Title: Levofloxacin-containing Therapies In Second Line Helicobacter Pylori Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Tai M.D., Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8C0201
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Proton pump inhibitor; Eradication
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Levofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential therapy (Experimental): Esomeprazole (Nexium)(40 mg) 1 tablet twice daily, amoxicillin (Amolin)(500 mg) 2 tablets twice daily for 5 days followed by esomeprazole (Nexium) (40 mg) twice daily, levofloxacin(Cravit)(500 mg), 1 tablet once daily and metronidazole (Flagyl)(250 mg) 2 tablets three times daily for 5 days
  Interventions: Drug: Nexium; Drug: Amolin; Drug: Cravit; Drug: Flagyl
- Triple therapy (Active Comparator): Esomeprazole (Nexium)(40 mg) 1 tablet twice daily; amoxicillin (Amolin)(500 mg) 2 tablets twice daily and levofloxacin(Cravit)(500 mg), 1 tablet once daily for 10 days
  Interventions: Drug: Nexium; Drug: Amolin; Drug: Cravit

INTERVENTIONS:
Drug: Nexium — Esomeprazole (Nexium)(40 mg) 1 tablet twice daily for 10 days in both arms
  Other Names: Esomeprazole
Drug: Amolin — Amoxicillin (Amolin)(500 mg) 2 tablets twice daily for the first 5 days in the Sequential arm; Amoxicillin (Amolin)(500 mg) 2 tablets twice daily for 10 days for triple therapy arm
  Other Names: Amoxicillin
Drug: Cravit — Levofloxacin(Cravit)(500 mg) 1 tablet once dialy for the last 5 days in the sequential arm and 1 tablets once daily for 10 days in the triple therapy arm
  Other Names: Levofloxacin
Drug: Flagyl — Metronidazole (Flagyl)(250 mg) 2 # tid for the last 5 days in the sequential arm
  Other Names: Metronidazole
  Arms: Sequential therapy

SUMMARY:
Asia Pacific Consensus states that levofloxacin-based triple therapy as an alternative second-line therapy after Helicobacter pylori (H. pylori) eradication failure when bismuth salts are not available. The investigators compare the efficacies of 10-day levofloxacin-based sequential therapy and 10-day triple therapy in the treatment for patients after failure of standard triple therapy and to determine what clinical and bacterial factors influencing the efficacy of salvage regimens.

DETAILED DESCRIPTION:
In this randomized-controlled trial , the investigator recruited participants with H pylori infection after failure of first line standard triple therapy. Using a computer-generated randomization sequence, the investigators randomly allocated patients to either 10-day levofloxacin-containing sequential (EALM, esomeprazole 40 mg b.d., amoxicillin 1 g b.d.for 5 days and followed by esomeprazole 40 mg b.d., levofloxacin 500 mg qd and metronidazole for 5 days) or 10-day levofloxacin-containing triple therapy (EAL, esomeprazole 40 mg b.d., amoxicillin 1 g b.d., and levofloxacin 500 mg qd) at a 1:1 ratio. The primary outcome was the eradication rate by intention-to-treat and per-protocol analyses.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H. pylori-infected participants, at least 18 years of age, with endoscopically proven peptic ulcer diseases or gastritis who failed first-line eradication therapies with standard triple regimens (PPI twice daily, 500 mg of clarithromycin twice daily and 1 g of amoxicillin twice daily)

Exclusion Criteria:

* Ingestion of antibiotics, bismuth, or proton-pump inhibitors within the prior 4 weeks
* Use of non-steroidal anti-inflammatory drugs within the prior 4 weeks
* Participants with allergic history to the medications used
* Participants with previous gastric surgery
* The coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Tai, M.D., Principal Investigator — Division of Hepatogastroenterology, Kaohsiung Chang Gung Memorial Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
mmmm

REFERENCES:
- [Result] Chuah SK, Tsay FW, Hsu PI, Wu DC. A new look at anti-Helicobacter pylori therapy. World J Gastroenterol. 2011 Sep 21;17(35):3971-5. doi: 10.3748/wjg.v17.i35.3971. PMID 22046084
- [Result] Tanaka M, Isogai E, Isogai H, Hayashi S, Hirose K, Kimura K, Sugiyama T, Sato K. Synergic effect of quinolone antibacterial agents and proton pump inhibitors on Helicobacter pylori. J Antimicrob Chemother. 2002 Jun;49(6):1039-40. doi: 10.1093/jac/dkf055. No abstract available. PMID 12039901
- [Result] Chuah SK, Tai WC, Lee CH, Liang CM, Hu TH. Quinolone-containing therapies in the eradication of Helicobacter pylori. Biomed Res Int. 2014;2014:151543. doi: 10.1155/2014/151543. Epub 2014 Aug 28. PMID 25243116
- [Result] Vakil N, Megraud F. Eradication therapy for Helicobacter pylori. Gastroenterology. 2007 Sep;133(3):985-1001. doi: 10.1053/j.gastro.2007.07.008. PMID 17854602
- [Result] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Result] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Result] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Result] Wu IT, Chuah SK, Lee CH, Liang CM, Lu LS, Kuo YH, Yen YH, Hu ML, Chou YP, Yang SC, Kuo CM, Kuo CH, Chien CC, Chiang YS, Chiou SS, Hu TH, Tai WC. Five-year sequential changes in secondary antibiotic resistance of Helicobacter pylori in Taiwan. World J Gastroenterol. 2015 Oct 7;21(37):10669-74. doi: 10.3748/wjg.v21.i37.10669. PMID 26457027
- [Derived] Chuah SK, Liang CM, Lee CH, Chiou SS, Chiu YC, Hu ML, Wu KL, Lu LS, Chou YP, Chang KC, Kuo CH, Kuo CM, Hu TH, Tai WC. A Randomized Control Trial Comparing 2 Levofloxacin-Containing Second-Line Therapies for Helicobacter pylori Eradication. Medicine (Baltimore). 2016 May;95(19):e3586. doi: 10.1097/MD.0000000000003586. PMID 27175657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 164 patients who had failed the H pylori eradication attempts using the standard triple therapy (proton pump inhibitor bid, clarithromycin 500 mg bid, amoxicillin 1 g bid × 7 days) were randomly assigned to either an sequential therapy group (EALM)(n = 82) or a 10-day levofloxacin-containing teriple therapy group (EAL)(n = 82).
Pre-assignment Details: We excluded those patients who had taken antibiotics, bismuth, proton-pump inhibitors, or non-steroidal anti-inflammatory drugs within the previous 4 weeks, were allergic to the medications used, had a history of previous gastric surgery or serious concomitant illness, or were currently pregnant.
Groups:
- Sequential Therapy: esomeprazole 40 mg bid and amoxicillin 1 g bid for 5 days, followed by esomeprazole 40 mg bid, levofloxacin 500 mg qd, and metronidazole 500 mg tid, for 5 days
- Triple Therapy: levofloxacin 500 mg qd, amoxicillin 1 g bid, and esomeprazole 40 mg bid
Period: Overall Study
Arm/Group | Sequential Therapy | Triple Therapy
Started | 82 (Started from 1st October 2013) | 82 (Started from 1st October 2013)
Completed | 81 (Completed on 30th September 2015) | 81 (Completed on 30th September 2015)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequential Therapy | Triple Therapy | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 68 | 138
  >=65 years | 12 | 14 | 26
Gender [Count of Participants; unit: Participants]
  Female | 46 | 42 | 88
  Male | 36 | 40 | 76
Region of Enrollment [Number; unit: participants]
  Taiwan | 82 | 82 | 164

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Eradication of H. Pylori
Description: Successful eradication of H. pylori is defined as (1) negative results of both rapid urease test and histology, or (2) a negative result of urea breath test at 4 weeks.
Time Frame: Negative results of H.pylori 4 weeks after eradication
Measure: Number (95% Confidence Interval); unit: percentage of eradication
Arm/Group | Sequential Therapy | Triple Therapy
Number analyzed (Participants) | 81 | 81
percentage of eradication | 91.4 [85.1 to 97.6] | 81.5 [72.8 to 90.1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Sequential Therapy | Triple Therapy
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 19/81 | 9/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequential Therapy (N=81) | Triple Therapy (N=81)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (General disorders) | 4 (4) | 1 (1)
Headache (General disorders) | 3 (3) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4)
Other (General disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes